CLINICAL TRIAL: NCT02394392
Title: Clinical Characteristics and Medication Satisfaction of Kanarb Tablet in Korean Hypertensive Patient: a Prospective, Cross-sectional and Open-label 8 Week Switching Study
Brief Title: Clinical Characteristics and Medication Satisfaction of Kanarb Tablet in Korean Hypertensive Patient(Kanarb-Hypertension Epidemiology Medication Satisfaction Study)
Acronym: K-HEMS
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-FMS-OB-401
Record Dates: First submitted 2015-03-10; First posted 2015-03-20 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension
Keywords: Medication satisfaction; Quality of life; Drug compliance
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1. Investigate the clinical characteristics, medication satisfaction and quality of life of anti-hypertensive drugs in Korean hypertensive patients
2. Observe the changes of medication satisfaction and compliance in patients after switchting to Fimasartan

ELIGIBILITY:
Inclusion Criteria:

Step1

* Over 20 years old
* Essential hypertensive patients who taking anti-hypertensive drugs during previous 1 month

Step2

* Patients does not taking Fimasartan
* Patient's medication satisfaction score under 4

Exclusion Criteria:

* Patients with secondary hypertension
* Patients with orthostatic hypotension who has sign and symptom
* Patients with known severe or malignancy retinopathy
* Patients with significant investigations; abnormal renal function
* Childbearing and breast-feeding women
* Patients with history of allergic reaction to any angiotensin II antagonist

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 14,000 hypertensive patients anticipated 30% of hypertensive patients who does not satisfied their anti-hypertensive drugs
Sampling Method: Non-Probability Sample
Enrollment: 12691 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
quality of life questionnaire for hypertension | up to 1 month
medication satisfaction questionnaire | up to 8 weeks

SECONDARY OUTCOMES:
Drug compliance questionnaire | up to 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Korea university Guro hospital, Seoul, South Korea

REFERENCES:
- [Derived] Oh DJ, Han SE, Jeong SH, Hong MS, Choe SC. Clinical characteristics and satisfaction with the fimasartan in Korean hypertensive patients: a prospective, cross-sectional and open-label, 8-week switching study (Kanarb-hypertension epidemiology medication satisfaction study; K-HEMS study). Clin Hypertens. 2018 Sep 1;24:10. doi: 10.1186/s40885-018-0096-2. eCollection 2018. PMID 30186623